CLINICAL TRIAL: NCT04153305
Title: European Registry for Myeloproliferative Neoplasms (MPNs) - Update of ERNEST Study
Acronym: ERNEST
Status: Completed | Type: Observational
Sponsor: FROM- Fondazione per la Ricerca Ospedale di Bergamo- ETS (Other)
Responsible Party: Sponsor
Other Study IDs: ERNEST - FROM/O1- 2019
Record Dates: First submitted 2019-11-04; First posted 2019-11-06 (Actual); Last update posted 2023-01-11 (Actual); Status verified 2023-01

CONDITIONS: Myelofibrosis
Keywords: survival; acute leukemia; second cancer; cardiovascular complication; update; disease management
MeSH Terms: conditions — Primary Myelofibrosis; Neoplasms, Second Primary

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: No

SUMMARY:
The Fondazione per la Ricerca Ospedale di Bergamo (FROM) decided to propose and promote the completion of ERNEST registry: the aim of the project is to obtain up-to-date estimates of clinical outcome of these patients in primary and secondary Myelofibrosis that have been included in the 'original' ERNEST study. The last was conducted between 2012 and beginning of 2015 including 1292 patients with Myelofibrosis, but it was interrupted in 2015 because of bankruptcy of the previous sponsor.

DETAILED DESCRIPTION:
Follow-up of patients already been registered in the ERNEST registry resulting alive and/or in active surveillance at November 2014 (Blood 2014 124:1849) will be updated retrospectively until December 2020. Data collection will be centralized at Fondazione per la Ricerca Ospedale di Bergamo (FROM), and performed by a web-based and Electronic Data Capture (EDC) system through ad hoc electronic case report forms (e-CRFs). The e-CRFs system will be pre-filled with pre-existing data collected from cases already entered in the registry. Information on therapies received and outcome events occurred (in term of death, evolution to acute leukemia, secondary cancer and cardiovascular complications) until December 2020 will be recorded by authorized participating investigators.

ELIGIBILITY:
Inclusion Criteria:

* previous registration in the ERNEST registry (2012 - 2014)
* diagnosis of MF performed between January 2001 and 2012 December
* Signed informed consent to continue participation in the registry

Exclusion Criteria:

None

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients aged 18 years old or more, with diagnosis of Primary Myelofibrosis (PMF), Post-Polycythemia Vera Myelofibrosis (PPV-MF) or Post-Essential Thrombocythemia Myelofibrosis (PET-MF) performed according WHO 2001 or WHO 2008, between 2001 and 2012.
Sampling Method: Probability Sample
Enrollment: 1010 (Actual)
Dates: Start 2019-10-08 (Actual); Primary Completion 2020-12-31 (Actual); Study Completion 2020-12-31 (Actual)

PRIMARY OUTCOMES:
Number of death | 18 years
  Overall Survival

SECONDARY OUTCOMES:
Number of patients with evolution to acute leukemia (AL) | 18 years
  Occurrence of AL from diagnosis to last observation
Number of patients with secondary tumor (ST) | 18 years
  Occurrence of ST from diagnosis to last observation
Number of patients with cardiovascular (CV) complications | 18 years
  Occurrence of events from diagnosis to last observation

CONTACTS AND LOCATIONS:
Overall Officials: Tiziano Barbui, MD, Study Chair — Fondazione per la Ricerca Ospedale di Bergamo
Locations (6):
- Italy (4):
  - AOU Careggi, Florence, FI
  - UOC Ematologia, ASST Papa Giovanni XXIII, Bergamo, Lombardy
  - Divisione Ematologia, Fondazione IRCCS Policlinico San Matteo, Pavia, Lombardy
  - U.O. Ematologia, Ospedale di Circolo e Fondazione Macchi Varese, Varese, Lombardy
- Hospital Clínic de Barcelona, Barcelona, Spain
- Center is Hematology Section, Uddevalla Hospital, Uddevalla, Sweden

IPD SHARING:
Plan to Share IPD: No